CLINICAL TRIAL: NCT06487403
Title: HN-BIO 02: A Phase II Randomized Study of the Effects of Delayed Elective Radiotherapy on Head and Neck MRI and Immune Response Biomarkers
Acronym: HN-Bio 02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-5510
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Integrated Boost Radiotherapy (Active Comparator): External beam radiotherapy 70Gy in 35 fractions to head and neck tumour and 56 Gy in 35 fraction to elective nodal regions. This will be given as single integrated boost or two-phase treatment at clinician discretion.
  Interventions: Radiation: Standard of care external beam radiotherapy (single integrated boost)
- Arm 2: Two Phase Radiotherapy (Active Comparator): Standard of care external beam radiotherapy 70 Gy in 35 fractions to head and neck with delayed 40 Gy in 20 fractions (HPV+ oropharynx) or 50 Gy/25 (all other disease) to elective nodal regions. This will be given as reversed two-phase treatment.
  Interventions: Radiation: Standard of care external beam radiotherapy (two-phase treatment)

INTERVENTIONS:
Radiation: Standard of care external beam radiotherapy (single integrated boost) — 70Gy in 35 fractions, 56 Gy in 35 fractions. Oral Pimonidazole 200 mg and 300 mg tablets.
  Arms: Arm 1: Integrated Boost Radiotherapy
Radiation: Standard of care external beam radiotherapy (two-phase treatment) — 70Gy in 35 fractions, delayed 40 Gy in 20 fractions or 50 Gy in 25 fractions. Oral Pimonidazole 200 mg and 300 mg tablets.
  Arms: Arm 2: Two Phase Radiotherapy

SUMMARY:
This is a single centre prospective exploratory study of effects of radiation therapy on biomarker development in patients with newly diagnosed (head and neck squamous cell carcinoma) HNSCC receiving curative therapy. This research is part 2 of the HN-BIO study.

DETAILED DESCRIPTION:
This study will recruit up to 40 patients planned to receive curative (chemo) radiotherapy for (head and neck squamous cell carcinoma) HNSCC with primary tumor and/or involved lymph node suitable for repeat biopsy in clinic. After being informed about the study and potential risks, patients giving written informed consent will be randomized to receive conventional radiotherapy (single integrated boost or conventional two-phase at clinician discretion) or reversed two-phase treatment with delayed irradiation of elective nodal volumes. Patients will not be informed of their randomization result.

Patients in both arms will undergo a baseline functional magnetic resonance imaging (fMRI) scan and within 72 hours, when possible, a biopsy of the primary tumor +/- lymph node will be performed in an out-patient clinic. If a suitable biopsy has been recently performed as part of diagnostic work up the baseline biopsy on study will be omitted when possible. In week 2 of radiotherapy, patients will have a second fMRI scan and a paired biopsy within 72 hours of the scan, where possible. A further optional biopsy and paired fMRI scan in week 4 will be considered for patients who are tolerating therapy without >G1 toxicities. 16-24 hours prior to each biopsy the patient will take oral pimonidazole. At the time of each biopsy a blood draw will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Histologically proven Head and Neck Squamous Cell carcinoma
* Primary or nodal disease > 3cm for biomarker imaging
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Planned for curative surgery or (chemo)radiotherapy
* Willingness to undergo repeat MRI imaging
* Able to receive and understand verbal and written information regarding study and able to -give written informed consent
* Adequate renal function: Calculated creatinine clearance >/= 30ml/min
* Be able to lie comfortably on back for 1 hour

Exclusion Criteria:

* As judged by investigator evidence of systemic disease that makes unsuitable for study
* Contra-indication for serial MRI scans
* Previous solid tumor treated within last 5 years
* Pregnancy
* History of gadolinium contrast allergy
* Non-reversible clotting abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Confirm feasibility of recruitment of HN patients for on treatment repeat biopsy of the primary tumor +/- neck nodes | 7 weeks
  Achieve a minimum recruitment rate of one patient per month.
Change in fMRI during radiotherapy | 7 weeks
  Study association of changes in fMRI and tissue biomarkers during radiotherapy. Assessed through hypoxic regions visible on imaging scans.
Assess changes in tumor microenvironment during differing radiotherapy scheduling via repeat biopsy. | 7 weeks
  Assess effect of varying radiotherapy treatment volumes on changes in tumor microenvironment via repeat biopsy before and during radiotherapy. Quantify effect of delayed treatment of dLN on dynamic changes tumor immune micro-environment and hypoxia status during radiotherapy. Perform exploratory analysis of study data correlating changes in tumor microenvironment and hypoxia status with disease response to therapy.

SECONDARY OUTCOMES:
Validate novel and established fMRI imaging as predictive and prognostic radiotherapy biomarkers for HNSCC | 7 weeks
  Correlate changes in TME and hypoxia with changes in fMRI on repeat assessment. Correlate fMRI characterized tumor with pathological post-operative specimen.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada